CLINICAL TRIAL: NCT04683601
Title: Generation of a Surgical Field at the Mid-lower Mediastinum for Thoracoscopic Esophagectomy in the Left Lateral Decubitus Position
Brief Title: Generation of a Surgical Field in the Left Lateral Decubitus Position
Status: Completed | Type: Observational
Sponsor: Shizuoka Cancer Center (Other)
Responsible Party: Principal Investigator, Kenjiro Ishii, Principal Investigator, Shizuoka Cancer Center
Other Study IDs: ShizuokaCC 2
Record Dates: First submitted 2020-12-14; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Esophageal Cancer; Thoracic Diseases
Keywords: Left decubitus position; Mid-lower mediastinum; Thoracoscopic esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms; Thoracic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Thoracoscopic esophagectomy in left decubitus — Making surgical field at thoracoscopic esophagectomy in left decubitus

SUMMARY:
The generation of a good surgical field at the mid-lower mediastinum during thoracoscopic esophagectomy in the left lateral decubitus position is often complicated. The investigators developed a simple and useful technique for surgical field generation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent thoracoscopic esophageal resection from April 2015 to December 2019 in our hospital.

Exclusion Criteria:

* patients who underwent open thoracotomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 154 patients underwent thoracoscopic esophagectomy in left decubitus position during that period.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Completion rate of thoracoscopic esophagectomy | During surgery
  The rate of completion of thoracic esophagectomy with our method for the generation of surgical field in mid-lower mediastinum.

IPD SHARING:
Plan to Share IPD: No